CLINICAL TRIAL: NCT04823663
Title: BoStOn SCientific Rhythm MAnagemenT REgiStry
Brief Title: BoStOn SCientific Rhythm MAnagemenT REgiStry (SOCRATES)
Acronym: SOCRATES
Status: Recruiting | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: SOCRATES - C2157; NCT04828811 (obsolete NCT alias)
Record Dates: First submitted 2021-03-18; First posted 2021-04-01 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases | interventions — Mutagenesis, Insertional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BSC Product Use: Subject fulfilling one of the following conditions:
  a. prospectively scheduled for a procedure involving i. use of a BSC EP Ablation product or BSC Capital Equipment product or ii. a BSC CRM product implant or b. retrospectively enrolled no more than 10 days after the index procedure and and all data necessary for appropriate reporting of all past visits is available and complete including i. the procedure where being diagnosed or treated with at least 3 separate BSC EP Ablation products/components or BSC Capital Equipment products/components or ii.the BSC CRM product implant.
  Interventions: Device: Implant; Procedure: Electrophysiologic procedure

INTERVENTIONS:
Device: Implant — In the scope of the CRM procedure and subsequent follow-up, the registry will provide information on the use of the Boston Scientific CRM products/components and combination of those products/components with competitor product(s) per hospital's standard of care.
Procedure: Electrophysiologic procedure — In the scope of the EP procedure and subsequent follow-up, the registry will provide information on the use of the Boston Scientific Electrophysiology products/components and capital equipment products and combination of those products/components with competitor product(s) per hospital's standard of care.

SUMMARY:
SOCRATES is part of Boston Scientific's (BSC) Post-market surveillance system. The implementation of such systems is mandatory per local regulations such as the Regulation '(EU) 2017/745 of the European Parliament and of the Council of 5 April 2017 on medical devices' or short Medical Device Regulation (MDR). The SOCRATES design is therefore based on the BSC's commitment as well as external regulatory requirements to proactively and systematically gather, record and analyze relevant data on the quality, performance and safety of devices throughout their entire lifetime.

DETAILED DESCRIPTION:
SOCRATES is a non-randomized, multisite, single-arm, open-label, global post-market observational data collection per standard of care. While generally of prospective design, a limited retrospective element is allowed for the inclusion of patients for a short period of 10 days after their index procedure.

SOCRATES intends to enroll a number of subjects that will support the analysis of all the individual Post Market Clinical Follow-Up (PMCF) Plans. An average of approximately 100 subjects per year and site on a continuous basis is expected but may vary depending on the needs of individual PMCF Plans. As long as SOCRATES is active, there is no upper limit to the total number of subjects that may be enrolled, and enrollment will be driven by the need to support sample sizes of individual PMCF plans for given products/product groupings supported by SOCRATES.

SOCRATES is designed to be a continuous effort after the data collection commences without a predefined closure timepoint. Data collection and enrollment may be stopped, restarted or finalized per Sponsor discretion.

The expected duration of SOCRATES participation for a subject is dependent on

* the specific lifetime of the device (e.g. the battery usage for pulse generators or continued active use of leads for CRM devices) or
* the necessary timeframe to adequately assess safety and performance of the device based on the residual risk assessed for each device in the associated PMCF plan. Timeframes might e.g. spread from 7 days to one year post procedure for EP. The maximum duration per enrolled subject will consequently vary.

For BSC implantable devices subjects are intended to be followed for the entire time of being implanted with a BSC device to allow data collection over the lifetime of the device(s) as required by applicable regulations. A maximum duration per enrolled subject is not defined, unless locally required. In case a local maximum duration is enforced subjects may be consented again and re-enrolled for continued participation if they are still in scope for SOCRATES. Sites shall ensure continuous data collection without any gaps in case a re-enrollment becomes applicable. Data sets for re-enrolled subjects will be handled as if the subject was continuously enrolled. This process will ensure to meet the requirement of MDR for device manufacturers to collect data over the lifetime of the devices.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is willing and capable of providing informed consent and/or to give approval to collect/store/process personal health information by the sponsor or such consent/approval is provided by a legally designated representative, if required by local law or regulation.
2. Subject is (one criterion must be fulfilled) a. prospectively scheduled for a procedure involving i. use of a BSC EP Ablation product or BSC Capital Equipment product or ii. a BSC CRM product implant or b. retrospectively enrolled no more than 10 days after the index procedure and all data necessary for appropriate reporting of all past visits is available and complete including i. the procedure where being diagnosed or treated with at least 3 separate BSC EP Ablation products/components or BSC Capital Equipment products/components or ii. the BSC CRM product implant.

Exclusion Criteria:

1. Subject is foreseen not to be followed at the enrolling center for at least 1 year after an implant procedure (CRM) or at least 1 month (EP).
2. Subject is receiving diagnosis or therapy by means of any product, that is not approved for commercial use at the time of implant/procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects will be recruited from the general patient population of the participating centers who are
  * receiving diagnosis or treatment using a BSC product in scope of SOCRATES and
  * fulfilling all inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 12500 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
System-related complication free rate | From Cardiac Rhythm Management (CRM) device implant on day 0 through follow-up up to 10 years; from electrophysiological (EP) procedure on day 0 through follow-up from 30 days up to 1 year
  Freedom from complications related to system
Rate of product related performance deficiencies per product or product group | CRM implant on day 0; EP procedure on day 0
  Performance of product/product group at implant/procedure
Rate of product related performance deficiencies per product or product group | CRM implant on day 0 through the implanted duration up to 10 years
  Performance of product/product group through the implanted duration

CONTACTS AND LOCATIONS:
Overall Officials: Eszter Pais, MD, Study Director — Boston Scientific Corporation
Locations (26):
- Belgium (2):
  - Universitair Ziekenhuis Brussel, Jette
  - CHU UCL Namur - Site Godinne, Yvoir
- Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec, Quebec, Canada
- France (5):
  - CHRU de Brest, Hôpital de la Cavale Blanche, Brest
  - CHRU de Clermont-Ferrand, Clermont-Ferrand
  - Hopital Saint Philibert, Lomme
  - CHG de Pau, Pau
  - CHU de Saint-Etienne, Saint-Etienne
- Germany (2):
  - Unfallkrankenhaus Berlin Marzahn, Berlin
  - Augusta Kranken Anstalt GmbH, Bochum
- Greece (2):
  - General Hospital of Athens "G. Gennimatas", Athens
  - Onassis Cardiac Surgery Center, Athens
- Mater Private Hospital, Dublin, Ireland
- Israel (3):
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourask Medical Center, Tel Aviv
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (4):
  - Policlinico di Modena, Modena
  - Policlinico Universitario Agostino Gemelli, Roma
  - Policlinico Casilino, Roma
  - Ospedale S.G. Calibita Fatebenefratelli - Isola Tiberina, Roma
- Spain (4):
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Nuestra Señora de La Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (2):
  - St. Bartholomew's Hospital, London
  - Manchester Heart Center, Manchester

IPD SHARING:
Plan to Share IPD: No